CLINICAL TRIAL: NCT06175741
Title: The Effect of Adding Morphine as an Adjuvant to Local Anesthetic in Erector Spinae Plane Block on Management of Acute Post Mastectomy Pain : A Randomized Controlled Trial
Brief Title: Adding Morphine to ESP Block in Management of Acute PMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadir atef, Principal invistigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESP block with morphine in PMP
Record Dates: First submitted 2023-11-30; First posted 2023-12-19 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Acute Post-mastectomy Pain Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): this group will receive erector spinae plane block only(bupivicaine)
  Interventions: Procedure: erector spinae plane block
- Interventional 3mg (Experimental): this group will receive erector spinae plane block (bupivicaine and 3mg morphine)
  Interventions: Procedure: erector spinae plane block
- Interventional 5mg (Experimental): this group will receive erector spinae plane block (bupivicaine and 5mg morphine)
  Interventions: Procedure: erector spinae plane block

INTERVENTIONS:
Procedure: erector spinae plane block — The ultrasound (US)-guided ESP block will be provided while the patient be in a seated position according to surgical site (right or left). Using high-frequency linear US transducer , the probe is placed in the longitudinal orientation lateral to thoracic third and six spinous processes ,then the trapezius muscle ,rhomboids major muscle and erector spinae muscle are identified and we will inject 20ml of 0.25% bupivacaine into interfacial plane below erector spinae muscle in one level (between T3and T6) ,alone in 1st group,with 3 mg morphine in 2nd group and 5 mg morphine in 3rd group

SUMMARY:
The aim of the study is to determine the efficacy of adding morphine in two doses (3mg, 5mg) to erector spinae plane block in relieving acute post mastectomy pain

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women requiring surgery . Breast surgeries is one of the most common type of surgery performed worldwide . Of these patients 30% to 50% will report moderate to severe acute pain. Pain if underestimated and untreated will affect patient's recovery , hemostasis, and lead to delayed discharge from PACU and increase length of hospital stay.Variety of local and regional anesthetic procedures which include local anesthetic infiltration , field block , intercostal nerve block , brachial plexus block and thoracic epidural anesthesia for breast surgery have considard as well established option to provide analgesia ,reduce post operative pain score , reduce opioid requirement , decrease post operative nausea and vomiting ,decrease pulmonary complication and duration of stay in PACU and specific to breast surgery there is also some evidence that regional anesthesia may help attenuate the surgical stress response and indirectly contribute to tumor inhibition by reducing opioid usage which has been implicated in immunosuppression and cancer progression. Pectoralis nerve block , serratus anterior nerve block and paravertebral nerve block are used for breast surgery analgesia . pectoralis nerve block and paravertebral block entrenched in clinical practice , and both of these techniques are shown to be effective as analgesic after breast surgery . However these techniques have many drawbacks . For example after performing the pectoralis nerve block the spread of the local anesthetic may interfere with surgical field . Paravertebral block can cause pneumothorax and epidural or intra thecal injection of the local anesthetic. Erector spinae plane block (ESPB) is a relatively new technique that was first described by Forero et Al in 2016 , they found that administration of local anesthetic below the erector spinae muscle produce extensive sensory block over the ipsilateral thorax . Forero et Al proposed that the injected local anesthetic spread anteriorly through the costo transverse foramen to its site of action at the origin of dorsal and ventral rami .Various adjuvants such as morphine , clonidine ,fentanyl, dexamethasone ,epinephrine ,and dexemedetomidine have been used with local anesthetic for improving and prolonging the postoperative analgesia with encouraging result . Morphine is a potent opioid analgesic widely used for treatment of severe pain. sedation scales assess the level of consciousness through behavioral observation and/ or stimulation of the patient. Ramsay sedation scale classifies level of awareness into six categories, this scale has multiple advantages :it is reproducible ,easy executed and has good applicability. This has made the scale the most widely used to assess level of sedation .Several rating scales have been developed to measure quality of recovery after surgery and anaesthesia, but the most extensively used after surgery is the QoR-40 scale,a40-item questionnaire that provide a global score and subscore across five dimension :patient support, comfort, emotion, physical independence, and pain.

ELIGIBILITY:
Inclusion Criteria:

* 1/female patients aged from 18 to 60 years.
* 2/ASA I -II
* 3/Surgery is modified radical mastectomy

Exclusion Criteria:

* 1/ASA more than II
* 2/Patients with known allergy to study drugs
* 3/Skin infection at site of needle puncture
* 4/Coagulopathy
* 5/Uncooperative patients

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
total morphine consumption | during 24 hours post operative
  . If the VAS score more than 3 rescue postoperative analgesia in the form of PCA morphine with initial bolus of 0.1mg/kg will be administered once the patient exhibit pain , followed by a 1 mg bolus with a locked period of 15 minutes when no background infusion will be permitted, total amount of morphine will be consumed be the patient will be recorded.

SECONDARY OUTCOMES:
Time of first analgesic request | 2,4,6,8,12,24 hours post operative
  time when the patient ask for analgesia post operative will be recorded
VAS at rest and movement | 2,4,6,8,12,24 hours post operative
  the visual analoge scale(VAS) which was scored from 0 to 10 where 0 = no pain and 10= the worst pain imaginable,
Mean blood pressure (MBP) | Pre operative,intra operative and post operative at 2,4,6,8,12,24 hours post operative
Number of participants with morphine side effects | 2,4,6,8,12,24 hours post operative
Ramsay sedation scale | 2,4,6,8,12,24 hours post operative
  Scale range from 1 (awake and alert) to 8 (unresponsive to external stimuli including pain)
Quality of recovery scale (QoR40) | at 24 hours post operative
  From 1 to 5, where 1=very poor and 5= excellent
Heart rate (HR) | Pre operative,intra operative and post operative at 2,4,6,8,12,24 hours post operative

CONTACTS AND LOCATIONS:
Overall Officials: shereen Mamdouh, Study Director — south Egypt cancer institute ,Assiut university

REFERENCES:
- [Background] Poleshuck EL, Katz J, Andrus CH, Hogan LA, Jung BF, Kulick DI, Dworkin RH. Risk factors for chronic pain following breast cancer surgery: a prospective study. J Pain. 2006 Sep;7(9):626-34. doi: 10.1016/j.jpain.2006.02.007. PMID 16942948
- [Background] Fecho K, Miller NR, Merritt SA, Klauber-Demore N, Hultman CS, Blau WS. Acute and persistent postoperative pain after breast surgery. Pain Med. 2009 May-Jun;10(4):708-15. doi: 10.1111/j.1526-4637.2009.00611.x. Epub 2009 Apr 22. PMID 19453965
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Weltz CR, Greengrass RA, Lyerly HK. Ambulatory surgical management of breast carcinoma using paravertebral block. Ann Surg. 1995 Jul;222(1):19-26. doi: 10.1097/00000658-199507000-00004. PMID 7618963
- [Background] Sekandarzad MW, van Zundert AAJ, Lirk PB, Doornebal CW, Hollmann MW. Perioperative Anesthesia Care and Tumor Progression. Anesth Analg. 2017 May;124(5):1697-1708. doi: 10.1213/ANE.0000000000001652. PMID 27828796
- [Background] Cali Cassi L, Biffoli F, Francesconi D, Petrella G, Buonomo O. Anesthesia and analgesia in breast surgery: the benefits of peripheral nerve block. Eur Rev Med Pharmacol Sci. 2017 Mar;21(6):1341-1345. PMID 28387892
- [Background] Zhao J, Han F, Yang Y, Li H, Li Z. Pectoral nerve block in anesthesia for modified radical mastectomy: A meta-analysis based on randomized controlled trials. Medicine (Baltimore). 2019 May;98(18):e15423. doi: 10.1097/MD.0000000000015423. PMID 31045802
- [Background] Bakshi SG, Karan N, Parmar V. Pectoralis block for breast surgery: A surgical concern? Indian J Anaesth. 2017 Oct;61(10):851-852. doi: 10.4103/ija.IJA_455_17. No abstract available. PMID 29242663
- [Background] Naja Z, Lonnqvist PA. Somatic paravertebral nerve blockade. Incidence of failed block and complications. Anaesthesia. 2001 Dec;56(12):1184-8. doi: 10.1046/j.1365-2044.2001.02084-2.x. PMID 11736777
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] El Mourad MB, Amer AF. Effects of adding dexamethasone or ketamine to bupivacaine for ultrasound-guided thoracic paravertebral block in patients undergoing modified radical mastectomy: A prospective randomized controlled study. Indian J Anaesth. 2018 Apr;62(4):285-291. doi: 10.4103/ija.IJA_791_17. PMID 29720754
- [Background] Hassan ME, Mahran E. Evaluation of the role of dexmedetomidine in improvement of the analgesic profile of thoracic paravertebral block in thoracic surgeries: A randomised prospective clinical trial. Indian J Anaesth. 2017 Oct;61(10):826-831. doi: 10.4103/ija.IJA_221_17. PMID 29242655
- [Background] Lozano-Diaz D, Valdivielso Serna A, Garrido Palomo R, Arias-Arias A, Tarraga Lopez PJ, Martinez Gutierrez A. Validation of the Ramsay scale for invasive procedures under deep sedation in pediatrics. Paediatr Anaesth. 2021 Oct;31(10):1097-1104. doi: 10.1111/pan.14248. Epub 2021 Jul 11. PMID 34173295
- [Background] Herrera FJ, Wong J, Chung F. A systematic review of postoperative recovery outcomes measurements after ambulatory surgery. Anesth Analg. 2007 Jul;105(1):63-9. doi: 10.1213/01.ane.0000265534.73169.95. PMID 17578958